CLINICAL TRIAL: NCT05869513
Title: The Effects of Krill Oil Supplementation on Adaptations in Muscle Strength, Function, Mass and Neuromuscular Function to a Pragmatic Home-based Resistance Exercise Intervention in Sedentary Older Adults: a Randomised Controlled Trial
Brief Title: Krill Oil and Resistance Exercise in Older Adults
Acronym: KOREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KOREA
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia
Keywords: Home exercise; Resistance exercise; Exercise; Krill oil; Muscle strength; Neuromuscular function; Physical function
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Plant Oils

STUDY DESIGN:
Intervention Model Description: 1:1 parallel group design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All supplements will be matched for taste and look
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vegetable oil + Resistance exercise (Placebo Comparator): 4g/day vegetable oil and home based resistance exercise for 16 weeks
  Interventions: Dietary Supplement: Vegetable oil; Other: Home-based resistance exercise
- Krill oil + Resistance exercise (Active Comparator): 4g/day krill oil and home based resistance exercise for 16 weeks
  Interventions: Dietary Supplement: Krill oil; Other: Home-based resistance exercise

INTERVENTIONS:
Dietary Supplement: Vegetable oil — Mixed vegetable oil
  Arms: Vegetable oil + Resistance exercise
Dietary Supplement: Krill oil — Superba Krill Oil
  Arms: Krill oil + Resistance exercise
Other: Home-based resistance exercise — Home based resistance band and body weight exercise

SUMMARY:
The aim of this study is to determine whether krill oil supplementation enhances effects of a pragmatic resistance exercise programme on adaptations in muscle strength, mass, function and neuromuscular function in sedentary older adults. Hypothesis - krill oil supplementation will enhance the beneficial effects of resistance exercise on muscle strength, function, mass and neuromuscular function in sedentary older adults.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 60 years
* scoring a low level of physical activity based on international physical activity questionnaire (not meeting the recommend physical activity which is at least 600 MET-min per week).

Exclusion Criteria:

* Diabetes
* severe cardiovascular disease
* seizure disorders
* uncontrolled hypertension (>150/90mmHg at baseline measurement)
* cancer or cancer that has been in remission <5 years
* ambulatory impairments which would limit ability to perform assessments of muscle function
* dementia
* taking medication known to affect muscle (e.g. steroids)
* have an implanted electronic device (e.g. pacemaker/defibrillator/insulin pump)
* on anticoagulant therapy
* allergies to seafood
* regular consumption of more than 1 portion of oily fish per week
* already taking fish or krill oil or other n3 PUFA supplements
* femoral neck fracture or other severe of hip or knee operations
* stroke
* Parkinson's disease
* COPD
* kidney disease
* hyperlipidaemia
* obesity
* osteoporosis.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Nueromuscular Junction (NMJ) transmission instability | Change from baseline to 16 weeks
  NMJ transmission instability will be measured by iEMG

SECONDARY OUTCOMES:
Knee extensor maximal torque | Change from baseline to 8 16 weeks
  Knee extensor maximal torque will be measured by a load cell
30s chair stand test | Change from baseline to 16 weeks
  measuring the functional abilities
Gait speed | Change from baseline to 16 weeks
  measuring the functional abilities
Force steadiness during submaximal isometric knee extensor contractions | Change from baseline to 16 weeks
  Steadiness of force whilst contracting
Red Blood Cell Omega-3 levels | Change from baseline to 16 weeks
Grip strength | Change from baseline to 16 weeks
  Grip strength will be measured by handgrip dynamometer
Muscle thickness | Change from baseline to 16 weeks
  Vastus Lateralis muscle thickness will be measured by ultrasound

OTHER OUTCOMES:
Step Time (sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Cycle Time (sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Step Length (cm) | Change from baseline to16 weeks
  Measured during a 4m walk using a gaitrite mat
Stride Length (cm) | Change from baseline to16 weeks
  Measured during a 4m walk using a gaitrite mat
H-H Base Support (cm) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Single Support (%GC) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Double Support (%GC) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Swing (%GC) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Stance (%GC) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Step/ Extremity Ratio | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Toe In / Out (deg) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Distance (cm) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Ambulation Time (sec) | Change from baseline to 16 weeks
Velocity (cm/sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Mean Normalized Velocity | Change from baseline to16 weeks
  Measured during a 4m walk using a gaitrite mat
Number of Steps | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Cadence (Steps/Min) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Step Time Differential (sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Step Length Differential (cm) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Cycle Time Differential (sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No